CLINICAL TRIAL: NCT05627752
Title: Docetaxel Alone or in Combination With Enzalutamide as First-line Treatment for Metastatic Castration Resistant Prostate Cancer Previously Treated With Abiraterone: a Single Center, Randomized, Open-label Study
Brief Title: Docetaxel Alone or in Combination With Enzalutamide for mCRPC Previously Treated With Abiraterone at mHSPC Stage
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhongnanH PCa
Record Dates: First submitted 2022-10-09; First posted 2022-11-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer; Castrate Resistant Prostate Cancer
Keywords: chemotherapy; Enzalutamide; Abiraterone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group of Combination (Experimental): Docetaxel plus Enzalutamide
  Interventions: Drug: Enzalutamide 40 MG; Drug: Docetaxel injection
- Group of Docetaxel (Placebo Comparator): Docetaxel plus placebo
  Interventions: Drug: Docetaxel injection

INTERVENTIONS:
Drug: Enzalutamide 40 MG — Adding Enzalutamide to Docetaxel chemotherapy
  Arms: Group of Combination
Drug: Docetaxel injection — Docetaxel chemotherapy

SUMMARY:
New androgen pathway targeting agents (ARTA), including Abiraterone acetate, Apalutamide and Enzalutamide, are approved and used in treatment of metastatic hormonal sensitive prostate cancer(mHSPC). However, the development of castration-resistance prostate cancer(CRPC) is only a matter of time. The use of sequential ARTAs in mCRPC showed limited benefit in retrospective series and prospective trials. Therefore this sequence should be avoided because of known cross resistance and the availability of chemotherapy and poly adenosine diphosphate-ribose polymerase(PARP) inhibitors (if a relevant mutation is present).

Recently, a randomized controlled trial(RCT), the ABIDO-SOGUG, indicated that compared with docetaxel, maintaining Abiraterone added to docetaxel in chemotherapy-naive patients who have experienced cancer progression to Abiraterone treatment could not improve radiographic progression-free survival or the other endpoints.However, another RCT, the PRESIDE trial, indicated that in patients who had progressed on Enzalutamide, continued Enzalutamide treatment in combination with docetaxel led to a significant improvement of PFS compared with placebo plus docetaxel.

The aims of this trial is to assess both the efficacy and safety of docetaxel in combination with Enzalutamide as first-line treatment in mCRPC patients progressed on Abiraterone.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma
* mCRPC
* Eastern Cooperative Oncology Group(ECOG) 0-1
* prior Abiraterone treatment

Exclusion Criteria:

* prior Enzalutamide or Docetaxel treatment

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | up to 6 months
  The time from the beginning of randomization to the first disease progression (that is, biochemical progression, tumor growth, or the discovery of new lesions) or death due to any reason.

SECONDARY OUTCOMES:
overall survival (OS) | up to 16 months
  Time from the beginning of randomization to death due to any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhonghua Yang, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol